CLINICAL TRIAL: NCT02406989
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1, Multiple-Ascending Dose Study of MS-553 in Healthy Volunteers
Brief Title: A Multiple-Ascending Dose Study of MS-553 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MingSight Pharmaceuticals Pty Limited (Industry)
Responsible Party: Sponsor
Organization: MingSight Pharmaceuticals, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-553-102
Record Dates: First submitted 2015-03-25; First posted 2015-04-02 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Safety and PK in Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MS-553 (Experimental): MS-553 oral tablet BID x 14 days
  Interventions: Drug: MS-553
- Placebo (Placebo Comparator): Placebo oral tablet BID x 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MS-553 — Study Drug
  Arms: MS-553
Drug: Placebo — Matching placebo to MS-553
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multiple-ascending dose study of MS-553 in healthy volunteers. Endpoints are safety, tolerability, and pharmacokinetics. Subjects are dosed for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* In good general health with BMI 18 to 32 kg/m2. Females must be nonpregnant, nonlactating, postmenopausal at least 2 years or surgically sterilized at least 6 months prior

Exclusion Criteria:

* History of skin rash, migraine, or clinically significant ocular diseases, conditions predisposing to QT prolongation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Adverse Events as a Measure of Safety and Tolerability | 14 days

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 14 days
Area under the Plasma Concentration versus Time Area under the Plasma Concentration versus Time Curve | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia